CLINICAL TRIAL: NCT04334525
Title: Promoting Healthier Eating Among Children in Restaurants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Associate Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003356; 1R01HD096748-01A1 (NIH)
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Diet, Healthy
Keywords: child; restaurant; nudging; repeated exposure; diet; health

STUDY DESIGN:
Intervention Model Description: A cluster-randomized design will be used. 6 locations of Anderson's, a regional quick-service restaurant in the Buffalo, New York, area will be paired based on income levels in the surrounding census tracts. A location from each pair will be randomized to each study group (intervention, control). Phased data collection will occur, with each pair of restaurants assigned to a cohort.
Masking Description: Participants know which kids' meals are being promoted based on the materials received in each study group -- e.g., placemats and frequent diner cards promoting two featured (healthier) meals vs. all kids' meals -- but the health focus and research questions are not stated explicitly to the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generic placemats and frequent diner cards (No Intervention): Participants will receive generic placemats listing all of the restaurant's kids' meals. Families will also receive a generic frequent diner card, which after purchasing (any) kids' meals across 6 occasions, makes them eligible for a free kids' meal of their choice during a predetermined redemption period. Corresponding signage will be displayed in the restaurant.
- Placemats and frequent diner cards promoting healthier meals (Experimental): Participants will receive placemats promoting healthier featured kids' meals and the opportunity to redeem their kids' meal token for a toy instead of dessert. Families will also receive a frequent diner card, which after purchasing one of the featured healthier kids' meals across 6 occasions, makes them eligible for a free kids' meal of their choice during a predetermined redemption period. Corresponding signage will be displayed in the restaurant.
  Interventions: Behavioral: Choice architecture + repeated exposure

INTERVENTIONS:
Behavioral: Choice architecture + repeated exposure — Participants will receive placemats promoting healthier featured kids' meals and the opportunity to redeem their kids' meal token for a toy instead of dessert. Families will also receive a frequent diner card, which after purchasing one of the featured healthier kids' meals across 6 occasions, makes them eligible for a free kids' meal of their choice during a predetermined redemption period.
  Arms: Placemats and frequent diner cards promoting healthier meals

SUMMARY:
Restaurants are normative eating contexts for many families. Restaurant meals tend to be higher in calories and lower in nutritional quality than those prepared at home. Targeting children's food selection in restaurants has the potential to improve diet quality, attenuate excess energy intake, and shape healthy habits. The objective of this study is to make healthier kids' meal options more appealing and easier to choose via an in-restaurant intervention that combines repeated exposure and choice architecture strategies. Six locations of a quick-service restaurant will be paired based on income levels in the surrounding census tracts. A location from each pair will be randomized to each study group (intervention, control). Recruitment and data collection will be conducted across 3 cohorts, with recruitment conducted during a family's regular visit. Study participation will involve 7 more visits to the location where the family was recruited, 6 of which will be during an exposure period of about 2 months. Families in intervention restaurants will receive placemats promoting healthier featured kids' meals. Participating families will also receive a frequent diner card which, after purchasing one of the featured healthier kids' meals across 6 occasions, makes them eligible for a free kids' meal of their choice during a predetermined redemption period. In the control group, generic placemats will be provided, and participating families will be provided with frequent diner cards that can be used for any kids' meals. The aims of this study are: (1) to test effects of a healthier kids' meal intervention on children's meal orders, and (2) to test effects of a healthier kids' meal intervention on children's dietary intake. It is hypothesized that (1a) children in the intervention restaurants will be more likely than controls to select one of the promoted healthier kids' meals at post-test, (1b) children in the intervention group will order fewer calories and desserts and less saturated fat, sodium, and sugar at post-test versus controls, (1c) the promoted healthier meals will make up a greater percentage of kids' meals ordered in intervention restaurants versus controls, based on sales data across the study period, and (2) compared to controls, children in the intervention group will consume fewer calories and less saturated fat, sodium, and sugar in the restaurant at post-test.

DETAILED DESCRIPTION:
Restaurants are normative eating contexts for many families. Restaurant meals tend to be higher in calories and lower in nutritional quality than those prepared at home. Targeting children's food selection in restaurants has the potential to improve diet quality, attenuate excess energy intake, and shape healthy habits. The objective of this study is to make healthier kids' meal options more appealing and easier to choose via an in-restaurant intervention that combines repeated exposure and choice architecture strategies.

Six locations of a quick-service restaurant will be paired based on income levels in the surrounding census tracts. A location from each pair will be randomized to each study group (intervention, control). Recruitment and data collection will be conducted across 3 cohorts. After recruitment, families will be asked to order and eat like they normally would. All participating families will then complete measures of children's orders, intake, and demographics. Then families will receive placemats and frequent diner cards. Families in intervention restaurants will receive placemats promoting healthier featured kids' meals. These families will also receive a frequent diner card, which after purchasing one of the featured healthier kids' meals across 6 occasions, makes them eligible for a free kids' meal of their choice during a predetermined redemption period. In the control group, generic placemats will be provided following baseline data collection, and families will also be provided with frequent diner cards that can be used for any kids' meals. During subsequent exposure periods, lasting about 2 months per cohort, families will return to the restaurant location where they were recruited on a weekly basis. Placemats will be available at the restaurant entrance, and corresponding signage will be displayed in the restaurant. In intervention restaurants, signs will advertise promoted meals and the option to select a toy in place of dessert. Participating children will be able to use their frequent diner card during this time to earn a free meal during the subsequent redemption period. Families will also be asked to complete a brief online survey once per week to monitor restaurant patronage. In each restaurant, study staff will conduct observations of a subsample of participating family and server interactions. Finally, post assessments will be completed during predetermined redemption periods, lasting about 3 months per cohort. Placemats and signage will still be available in restaurants during this time. Study staff will collect the frequent diner cards and ask families to order and eat like they normally would and to not throw out any food or leftovers. Families will be able to redeem any earned free kids' meals during this time. When the family is done eating, study staff will approach the table to administer study measures assessing orders, perspectives on the meal, and intake. Finally, families will also be prompted to complete an online dietary recall (ASA24) after their post assessment.

The specific aims of this study are: (1) to test effects of a healthier kids' meal intervention on children's meal orders, and (2) to test effects of a healthier kids' meal intervention on children's dietary intake. It is hypothesized that (1a) children in the intervention restaurants will be more likely than controls to select one of the promoted healthier kids' meals at post-test, (1b) children in the intervention group will order fewer calories and desserts and less saturated fat, sodium, and sugar at post-test versus controls, (1c) the promoted healthier meals will make up a greater percentage of kids' meals ordered in intervention restaurants versus controls, based on sales data across the study period, and (2) compared to controls, children in the intervention group will consume fewer calories and less saturated fat, sodium, and sugar in the restaurant at post-test.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English (parent/guardian & child)
* 18 years or older (parent/ guardian)
* Between the ages of 4-8 years (child)
* Eats food from restaurants at least 2-3 times per month (child)
* Does not have allergies that preclude safe participation in the study (child)
* Eating a meal in the restaurant at the time of recruitment/baseline assessment
* Did not participate in pilot phase of this study, which involved taste tests of possible healthier meal options at the same restaurant chain

Exclusion Criteria:

* Is under 18 years of age (parent/ guardian)
* Does not have a child in the range of 4-8 years
* Does not speak English fluently (parent/guardian & child)
* Does not eat food from a restaurant at least 2-3 times per month (child)
* Has food allergies that preclude safe participation in the study (child)
* Not eating a meal in the restaurant at recruitment/baseline
* Participated in pilot phase of this study, which involved taste tests of possible healthier meal options at the same restaurant chain

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 241 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-24 (Actual)

PRIMARY OUTCOMES:
Meal type ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Whether a healthier children's meal or other children's meal was ordered
Change in meal type ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Whether a healthier children's meal or other children's meal was ordered
Total calories ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total calories ordered
Child in total calories ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total calories ordered
Total saturated fat ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total saturated fat ordered.
Change in total saturated fat ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total saturated fat ordered.
Total sugar ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total sugar ordered.
Change in total sugar ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total sugar ordered.
Total sodium ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total sodium ordered.
Change in total sodium ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Nutrition information provided by the restaurant will be combined with parent report of children's orders to calculate total sodium ordered.
Dessert ordered for child in restaurant | Post-test (about 4 months after recruitment)
  Whether or not a dessert was ordered
Change in dessert ordered for child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Whether or not a dessert was ordered

SECONDARY OUTCOMES:
Calories consumed at restaurant by child in restaurant | Post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total calories in the full item to calculate calories consumed.
Changes in calories consumed at restaurant by child in restaurant | Baseline, post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total calories in the full item to calculate calories consumed.
Saturated fat consumed at restaurant by child in restaurant | Post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total saturated fat in the full item to calculate saturated fat consumed.
Changes in saturated fat consumed at restaurant by child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total saturated fat in the full item to calculate saturated fat consumed.
Sugar consumed at restaurant by child in restaurant | Post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total sugar in the full item to calculate sugar consumed.
Changes in sugar consumed at restaurant by child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total sugar in the full item to calculate sugar consumed.
Sodium consumed at restaurant by child in restaurant | Post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total sodium in the full item to calculate sodium consumed.
Changes in sodium consumed at restaurant by child in restaurant | Baseline, midpoints 1-6 (weekly assessments about 2 months after recruitment), post-test (about 4 months after recruitment)
  Children's dietary intake will be measured using plate waste methodology. Grams consumed will be converted to percentages using total grams from pre-weights, and these percentages will be multiplied by the total sodium in the full item to calculate sodium consumed.

OTHER OUTCOMES:
Healthier children's meals ordered at aggregate level | Through study completion, an average of 3 years
  Aggregated sales data from the restaurant will be collected to monitor sales of healthier kids' meals across all patrons in Anderson's restaurants by study group during the study period.
Healthier children's meals ordered at aggregate level | Exposure period (about 2 months after participant recruitment)
  Aggregated sales data from the restaurant will be collected to monitor sales of healthier kids' meals across all patrons in Anderson's restaurants by study group during the exposure period.
Healthier children's meals ordered at aggregate level | Post-test (about 4 months after participant recruitment)
  Aggregated sales data from the restaurant will be collected to monitor sales of healthier kids' meals across all patrons in Anderson's restaurants by study group during the redemption/post-test period.
Changes in kids' meals ordered at aggregate level | 1 year prior to baseline through study completion, an average of 4 years
  Aggregated sales data from the restaurant will be collected to monitor sales of kids' meals across all patrons in Anderson's restaurants during the recruitment/baseline, exposure, and redemption/post-test periods and parallel time points one year prior.
Total daily calories consumed by child | Post-test (about 4 months after recruitment)
  Parents will report children's daily dietary intake using the Automated Self-administered 24-hour Dietary Assessment Tool (ASA24) the day after the in-restaurant part of the post-test assessment.
Total saturated fat consumed by child | Post-test (about 4 months after recruitment)
  Parents will report children's daily dietary intake using the Automated Self-administered 24-hour Dietary Assessment Tool (ASA24) the day after the in-restaurant part of the post-test assessment.
Total sugar consumed by child | Post-test (about 4 months after recruitment)
  Parents will report children's daily dietary intake using the Automated Self-administered 24-hour Dietary Assessment Tool (ASA24) the day after the in-restaurant part of the post-test assessment.
Total sodium consumed by child | Post-test (about 4 months after recruitment)
  Parents will report children's daily dietary intake using the Automated Self-administered 24-hour Dietary Assessment Tool (ASA24) the day after the in-restaurant part of the post-test assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Anzman-Frasca, PhD, Principal Investigator — University at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anzman-Frasca S, Tauriello S, Epstein L, Ferrante MJ, Gampp A, Goldsmith J, Haines J, Leone LA, Paluch R. Promoting Healthier Meal Selection and Intake Among Children in Restaurants: Protocol for a Cluster-Randomized Trial. JMIR Res Protoc. 2025 Oct 10;14:e73618. doi: 10.2196/73618. PMID 41072006